CLINICAL TRIAL: NCT04954222
Title: Tracking the Recovery of Respiratory Physiology in COVID-19 Patients a Pilot Study
Brief Title: Recovery of Respiratory System in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Courtney M. Wheatley, Co-Principal Investigator, Mayo Clinic
Other Study IDs: 21-001028
Record Dates: First submitted 2021-06-30; First posted 2021-07-08 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19 long haulers: Individuals that have been diagnosed with COVID19 and continue to have lingering symptoms associated with COVID19
- COVID19 no residual symptoms: Individuals that have been diagnosed with COVID19 and do not have lingering symptoms that are associated with COVID19

SUMMARY:
The purpose of this study is to determine the effects of the clinical course of treatment as well as long-term symptoms of COVID-19 on respiratory function, exercise capacity, and quality of life.

DETAILED DESCRIPTION:
This study will be completed over 4 sessions at the Mayo Clinic at either the Scottsdale Arizona or Rochester Minnesota locations. You will be asked to complete a series of questionnaires, lung function tests, and exercise tests at two time points: ≥ 28 days post diagnosis and 4-6 months after the first laboratory visit. All visits will take approximately 2 hours. During visits 1 and 3 a series of questionnaires as well as breathing tests, and an exercise test will be completed on a stationary bike. You will also be asked to breathe a gas mixture out of a bag to obtain measures of gas movement and sensitivity. During visits 2 and 4 you will complete an exercise test on a stationary bike to measure changes from the previous exercise test and a chest scan.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented positive qRT-PCR for SARS-CoV-2 confirming prior COVID-19 diagnosis
* At least 18 years of age.
* Female subjects must not be pregnant or trying to become pregnant during the duration of study participation.
* No known plans to move out of the state, or become unable to return to one of the Mayo Clinic sites for follow-up testing.
* Must be able to provide clear informed written consent.

Exclusion Criteria:

* Individuals with pacemakers or other implantable devices that will make interpreting a CT scan challenging.
* Individuals with major limitations to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female participants that have tested positive for COVID-19 within 28 or more days will be recruited for this study. Individuals with or without continuing symptoms of COVID-19 can participate.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Change in diffusion capacity of the lungs | through study completion, an average of 5 months
  change in diffusing capacity of the lungs for carbon monoxide and its components
Change in airway morphology | through study completion, an average of 5 months
  CT assessment of airway diameter and thickness
change basic spirometry | through study completion, an average of 5 months
  Measurement of basic lung function using forced vital capacity (FVC), slow vital capacity (SVC),
  forced expiratory volume at one second (FEV1), maximal inspiratory pressure (MIPS), maximal expiratory pressure (MEPS), exhaled nitric oxide (ExNO), forced oscillation technique (FOT), overnight pulse oximetry
Change in peak aerobic capacity | through study completion, an average of 5 months
  Change in examine post exertional malaise
Presence of post-exertional malaise | through study completion, an average of 5 months
  Evaluation of change in performance on maximal exercise test over two days to identify presence of post-exertional malaise
Change in symptoms | through study completion, an average of 5 months
  St. George's respiratory Questionnaire scoring of pulmonary symptoms. Scores range from 0 to 100, with higher scores indicating more limitations.
change in quality of life | through study completion, an average of 5 months
  SF-36 questionnaire assessment of physical and mental health. Two scores one for physical functioning and one for mental functioning. Scores range from 0-100 with a higher score indicating better health

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Johnson, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials